| Patient: Mahnoor Age: 27 Gender: Female |
|---|
| Case No: 155 / 24 |
| Doctor: Dr. Aatikah |
| parent/guardian of this child, declare that the purpose of this research has been explained to me by Dr. Aatkah I have been given the opportunity to ask questions and clear any queries I have about participating |
| in this research. |
| I have been ensured that the participation of in this study will not harm or reduce the quality of my |
| treatment. |
| I voluntarily participate in this research. |
| Parent/guardian signature: |
| Researcher Signature: <u>Aatikah</u> |
| Date: 19/9/24 |

## Informed Consent Form for Comparison Of Alignment Efficiency Of Steel Vs Elastomeric Ligatures In Lower

## Anterior Teeth: A Randomized Clinical Trial.

| Patient: | _ |
|---|---|
| Age: | _ |
| Gender: | _ |
| Case No: | _ |
| Doctor: | _ |
| I, Mr./Mrs | , parent/guardian of this child, declare |
| that the purpose of this research h | nas been explained to me by Dr |
| I have been given the opportunit | y to ask questions and clear any queries I have about participating |
| in this research. | |
| I have been ensured that the part | ticipation of in this study will not harm or reduce the quality of my |
| treatment. | |
| I voluntarily participate in this res | earch. |
| Date: | |
| | <del>_</del> |
| Researcher Signature: | |

